CLINICAL TRIAL: NCT07187843
Title: Study of the Progression of Axial and Cognitive Symptoms and Biomarkers of Neurodegeneration in Patients With Parkinson's Disease Divided Into Brain-first and Body-first Phenotypes
Brief Title: Study of Axial and Cognitive Symptoms and Biomarkers of Neurodegeneration in Brain-first and Body-first PD
Acronym: BRABOAXPD
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 350/2024/OSS/AUSLRE
Record Dates: First submitted 2025-09-03; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Parkinsonian Disorders; Brain Disease; Basal Ganglia Diseases; Synucleinopathies
Keywords: Neurodegenerative Diseases; Nervous System Diseases; Movement Disorders; biomarker; neuroinflammation; brain-first; body-first; axial symptoms
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Brain Diseases; Basal Ganglia Diseases; Synucleinopathies; Neurodegenerative Diseases; Nervous System Diseases; Movement Disorders; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Parkinson's Disease (Brain-First phenotype): Patients with early-stage Parkinson's disease without REM sleep behavior disorder (RBD), consistent with a Brain-First phenotype. These patients typically show early central dopaminergic deficits followed by peripheral involvement.
  Interventions: Other: Clinical assessments; Other: Phenotypic classification
- Early Parkinson's Disease (Body-First phenotype): Patients with early-stage Parkinson's disease with REM sleep behavior disorder (RBD) before or at motor onset, consistent with a Body-First phenotype. These patients are expected to show early peripheral involvement (e.g., cardiac MIBG denervation) preceding central dopaminergic loss.
  Interventions: Other: Clinical assessments; Other: Phenotypic classification

INTERVENTIONS:
Other: Clinical assessments — standardized neurological examination, motor and non-motor symptom scales, cognitive testing, and autonomic symptom questionnaires.
Other: Phenotypic classification — patients will be stratified into Brain-First and Body-First phenotypes based on the presence of RBD and instrumental findings.

SUMMARY:
This observational study aims to systematically characterize a cohort of patients with early-stage Parkinson's disease (PD) attending the Movement Disorders Center of AUSL-IRCCS Reggio Emilia, Italy. PD is the second most common neurodegenerative disorder, affecting about 1% of individuals over 60 years of age. The project will explore clinical and biological differences between the recently proposed "Brain-First" and "Body-First" phenotypes of PD. Patients will undergo detailed clinical evaluation, neuroimaging, and biomarker assessments (including neurodegeneration and neuroinflammation markers). Particular attention will be given to the progression of axial and cognitive symptoms, which represent major contributors to disability.

Findings from this study are expected to improve early patient stratification, clarify disease mechanisms, and support the development of precision medicine strategies and future disease-modifying therapies.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder after Alzheimer's disease, affecting up to 1% of individuals over the age of 60. While treatment remains symptomatic and no disease-modifying therapies are currently available, increasing research efforts are focusing on precision medicine approaches and the identification of disease subtypes that may guide prognosis and therapy.

Historically, PD patients have been classified according to motor (tremor-dominant, akinetic-rigid, axial) and non-motor features (sleep disturbances, autonomic dysfunction, mood disorders, fatigue, pain, weight loss, cognitive impairment). Genetic classifications have also been introduced, with approximately 10-15% of patients carrying mutations such as GBA or LRRK2, which are associated with earlier onset and potentially more aggressive disease.

In the early 2000s, Braak and colleagues proposed a neuropathological staging system in which α-synuclein pathology progresses in a stereotypical pattern from peripheral to central structures. More recent clinical and pathological evidence, however, has challenged this model and led to the proposal of two distinct subtypes: Brain-First and Body-First. In Brain-First PD, pathology begins in the central nervous system and spreads to the autonomic system; in Body-First PD, pathology originates in peripheral structures such as the enteric nervous system, propagating rostrally to involve the brain. REM sleep behavior disorder (RBD) has emerged as a clinical marker of the Body-First subtype.

This study will systematically characterize patients with early-stage PD, combining detailed clinical evaluation with instrumental assessments including neuroimaging and blood-based biomarkers. In particular, the project will investigate whether Brain-First and Body-First phenotypes differ in terms of:

* Clinical progression (with focus on axial and cognitive symptoms).
* Neurodegeneration biomarkers, including neurofilament light chain.
* Neuroinflammation markers, such as immune responses to α-synuclein, interferon-gamma, and interleukin-5.

The overarching goal is to identify biological and clinical markers that distinguish PD subtypes, improve early stratification, and support the development of targeted, disease-modifying therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD according to the MDS Clinical Diagnostic Criteria for Parkinson's Disease divided into brain-first and body-first phenotypes, based on the presence or absence of a REM sleep behavior disorder diagnosed using ambulatory polysomnography methods according to the criteria of the International Classification of Sleep Disorders (ICSD-3) criteria and on data from SPECT with DATSCAN and myocardial innervation scintigraphy [123I-MIBG].
* Free and informed consent expressed by the participant.
* At least 18 years of age.

Exclusion Criteria:

* Inability to express free and informed consent.
* Patient with a doubtful diagnosis.
* Participant under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with early-stage Parkinson's disease (PD) attending the Movement Disorders Center of AUSL-IRCCS Reggio Emilia. Eligible participants will be adults diagnosed with PD according to international clinical criteria, in the initial stages of the disease, and not yet affected by major motor or cognitive disability. Patients will be characterized from both a clinical and instrumental perspective, including motor and non-motor symptoms, genetic background, and biomarkers of neurodegeneration and neuroinflammation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the progression of axial symptoms | baseline, 12, 24, 36,48, 60 months
  Differences in quantitative parameters of gait (phase duration, root mean square of the acceleration of the trunk in x, y, z axes) assessed through the instrumented Timed Up and Go test (phases considered: overall iTUG, sit-to-stand, sitting, first turn, second turn, walking forward, return gait) between the brain-first and body-first groups at diagnosis and at subsequent annual follow-up visits (5-year follow-up) in OFF-medication and ON-Medication (both in single and dual task) conditions.
Risk of falling in the two subgroups, brain-first and body-first | baseline, 12, 24, 36,48, 60 months
  Assessment of possible differences in scores obtained on the Walking Handicap Scale (WHS) at baseline and at subsequent annual follow-up visits (5-year follow-up). The Walking Handicap Scale (WHS) measures walking ability and community mobility across six levels, from limited physiological walking to unrestricted social ambulation. Possible scores range from 1 (most limited walking ability) to 6 (fully independent walking in social environments); higher scores indicate better walking function.
Risk of falling in the two subgroups, brain-first and body-first | baseline, 12, 24, 36,48, 60 months
  Assessment of possible differences in scores obtained on the Hendrich II Fall Risk Model (HIIFRM) at baseline and at subsequent annual follow-up visits (5-year follow-up). The Hendrich II Fall Risk Model (HIIFRM) assesses fall risk using clinical variables including confusion/disorientation/impulsivity, symptomatic depression, altered elimination, dizziness, gender, use of antiepileptics or benzodiazepines, and performance on the "Get-Up-and-Go" test. Possible total scores range from 0 (lowest fall risk) upwards (commonly up to about 16 depending on version); higher scores indicate greater fall risk.
Assessment of the progression of axial symptoms | baseline, 12, 24, 36,48, 60 months
  Differences in quantitative parameters of balance (center of pressure mean position referred to the mid-point of the heels, area of the 95% confidence ellipse, sway mean velocities and root mean square displacements in the antero-posterior and medio-lateral directions) assessed through a static posturography test (with eyes open) between the brain-first and body-first groups at diagnosis and at subsequent annual follow-up visits (5-year follow-up) in OFF-medication and ON-Medication (both in single and dual task) conditions.

SECONDARY OUTCOMES:
Assessment of disease progression | baseline, 12, 24, 36,48, 60 months
  Assessment of the differences in the MDS-UPDRS total scores (part I, II, III, IV) and subscores (tremor, bradykinesia, rigidity, postural instability and gait difficulty, gait, dyskinesia and fluctuations subscores) in the study population at baseline and at subsequent annual follow-up visits (5-year follow-up).
Assessment of the progression of neurodegeneration and inflammatory biomarkers (neurofilaments, interferon-γ, cell-mediated anti-α-synuclein responses). | baseline, 12, 24, 36,48, 60 months
  Assessment of the differences in neurodegeneration and inflammatory biomarkers (neurofilaments, interferon-γ, cell-mediated anti-α-synuclein responses) in a subset of 50 patients in the study population. Analysis of differences in neurofilament levels and cell-mediated responses at baseline and at subsequent annual follow-up visits (5-year follow-up).
Brain MRI: analysis of differences in qualitative and quantitative parameters extrapolated at diagnosis. | 24 months
  Assessment of quantitative differences in the degree of cortical and subcortical atrophy (volumetric automated segmentation of cerebral regions with the Quibim Precision software® quantified as % of intracranial volume) in the study population assessed through volumetric 1.5 Tesla brain MRI at baseline.
Baseline Assessment of Nigrostriatal and Myocardial Denervation. | 24 months
  Semiquantitative assessment (heart to mediastinum ratio [H/M]) of differences in myocardial denervation in the study population through cardiac 123I-MIBG scintigraphy (early and delayed imaging)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Piancino MG, Farina D, Talpone F, Merlo A, Bracco P. Muscular activation during reverse and non-reverse chewing cycles in unilateral posterior crossbite. Eur J Oral Sci. 2009 Apr;117(2):122-8. doi: 10.1111/j.1600-0722.2008.00601.x. PMID 19320720
- [Background] Cavallieri F, Gessani A, Merlo A, Campanini I, Budriesi C, Fioravanti V, Di Rauso G, Feletti A, Damiano B, Scaltriti S, Guagnano N, Bardi E, Corni MG, Antonelli F, Cavalleri F, Molinari MA, Contardi S, Menozzi E, Puzzolante A, Vannozzi G, Bergamini E, Pavesi G, Fraix V, Meoni S, Fraternali A, Versari A, Lusuardi M, Biagini G, Pinto S, Moro E, Valzania F. Interplay between speech and gait variables in Parkinson's disease patients treated with subthalamic nucleus deep brain stimulation: A long-term instrumental assessment. Eur J Neurol. 2023 Jul;30(7):1963-1972. doi: 10.1111/ene.15803. Epub 2023 Apr 10. PMID 36971736
- [Background] Merlo A, Zemp D, Zanda E, Rocchi S, Meroni F, Tettamanti M, Recchia A, Lucca U, Quadri P. Postural stability and history of falls in cognitively able older adults: the Canton Ticino study. Gait Posture. 2012 Sep;36(4):662-6. doi: 10.1016/j.gaitpost.2012.06.016. Epub 2012 Jul 24. PMID 22832469
- [Background] Horsager J, Knudsen K, Sommerauer M. Clinical and imaging evidence of brain-first and body-first Parkinson's disease. Neurobiol Dis. 2022 Mar;164:105626. doi: 10.1016/j.nbd.2022.105626. Epub 2022 Jan 11. PMID 35031485
- [Background] Horsager J, Andersen KB, Knudsen K, Skjaerbaek C, Fedorova TD, Okkels N, Schaeffer E, Bonkat SK, Geday J, Otto M, Sommerauer M, Danielsen EH, Bech E, Kraft J, Munk OL, Hansen SD, Pavese N, Goder R, Brooks DJ, Berg D, Borghammer P. Brain-first versus body-first Parkinson's disease: a multimodal imaging case-control study. Brain. 2020 Oct 1;143(10):3077-3088. doi: 10.1093/brain/awaa238. PMID 32830221
- [Background] Bohnen NI, Postuma RB. Body-first versus brain-first biological subtyping of Parkinson's disease. Brain. 2020 Oct 1;143(10):2871-2873. doi: 10.1093/brain/awaa293. PMID 33103732